CLINICAL TRIAL: NCT01765946
Title: Effects of Metformin on Longevity Gene Expression and Inflammation and Prediabetic Individuals. A Placebo-controlled Trial
Brief Title: Metformin and Longevity Genes in Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Angelo Avogaro, Full professor of Endocrinology and Metabolism, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MetAge
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Insulin Resistance; Prediabetes; Aging; Inflammation
Keywords: Insulin resistance; Prediabetes; Longevity genes; Inflammation; Metformin
MeSH Terms: conditions — Insulin Resistance; Prediabetic State; Inflammation | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin tablets 500 mg tid for 2 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tables tid for 2 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metformin — Metformin tablets 500 mg tris in die (tid)
  Other Names: Glucophage
  Arms: Metformin
Drug: placebo
  Arms: Placebo

SUMMARY:
Pre-diabetes, a condition characterized by hyperglycaemia, is associated with increased cardiovascular risk and reduced life expectancy, as compared to the general population. AMP-activated protein kinase (AMPK) is an enzyme that plays a key role in cellular energy homeostasis and metabolism, and recently it has been demonstrated that AMPK regulates aging pathways, as well. AMPK is susceptible to modulation through pharmacologic (e.g. metformin) and non-pharmacologic (e.g. physical exercise) interventions. This clinical trial aims to describe the effects of the AMPK pathway on longevity genes and inflammation in the setting of pre-diabetes in vivo and in vitro. To this end, the investigators will compare treatment with metformin (500 mg t.i.d) for 2 months, versus placebo in pre-diabetic subjects. The investigators will assess expression of longevity genes SIRT1, p66Shc, p53 and mTOR in peripheral blood mononuclear cells (PBMCs) ex vivo. The investigators will evaluate monocyte polarization by flow cytometry, according to the expression of surface antigens (CD68, CCR2, CD163, CD206, CX3CR1) to determine the prevalence of pro- or anti-inflammatory cells. Inflammatory cytokines (TNF-alpha, MCP-1, IL-1, IL-6, IL-10, CCL12) will also be determined. In the in vitro study the investigators will evaluate the effects of AMPK activation or inhibition on longevity gene and protein expression.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes, defined as IFG (fasting glucose between 100 and 125 mg/dl) or IGT (2h post-oral glucose load (75g) between 140 and 199 mg/dl);
* Age 40-75 years;
* Both genders.

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus;
* Pregnancy, lactation;
* Acute, chronic or inflammatory diseases;
* Neoplasms;
* Immunological diseases, organ transplantation, steroid therapy;
* Uncontrolled arterial hypertension (systolic pressure > 180 mmHg or diastolic > 120 mmHg);
* Recent(within 3 months) surgical intervention or cardiovascular accidents;
* Known allergy to metformin.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Longevity gene expression | 2 month after treatment
  Change in the expression of longevity genes Sirtuin-1, p66Shc, mTor, p53 in peripheral blood mononuclear cells (PBMC)

SECONDARY OUTCOMES:
Insulin sensitivity | 2 months after treatment
  A dynamic measure of insulin sensitivity (Si) from the frequently sampled OGTT
Monocyte polarization status | 2 months after treatment
  Polarization of circulating monocytes in M1 (CD68+CCR2+) and M2 (CX3CR1+CD163+/CD206+)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Avogaro, M.D. Ph.D., Principal Investigator — University of Padova
Locations (1):
- University Hospital Diabetes Outpatient Clinic, Padua, Italy, Italy

REFERENCES:
- [Derived] de Kreutzenberg SV, Ceolotto G, Cattelan A, Pagnin E, Mazzucato M, Garagnani P, Borelli V, Bacalini MG, Franceschi C, Fadini GP, Avogaro A. Metformin improves putative longevity effectors in peripheral mononuclear cells from subjects with prediabetes. A randomized controlled trial. Nutr Metab Cardiovasc Dis. 2015 Jul;25(7):686-93. doi: 10.1016/j.numecd.2015.03.007. Epub 2015 Mar 24. PMID 25921843